**Title**: Medical-legal partnerships to prevent evictions and homelessness among veterans

NCT Number: NCT04924088

**IRB** approval date: May 10, 2023

### RESEARCH CONSENT FORM

# **VA Connecticut Healthcare System**

| Subject Name: | Date: |
|---|---|
| Title of Study: Medical-legal partnerships to prevent evictions and homelessness among veterans | |
| Principal Investigator: Marc Rosen, M.D. | Version Date: v.04/05/2023 |

#### **RESEARCH SUMMARY**

You are invited to take part in a research study because you are a Veteran looking for legal help with a problem related to your housing. This study is funded by the VA Office of Rehabilitation Research and Development (RR&D). Before you decide to take part, it is important for you to know why the research is being done and what it will involve. This initial summary is to give you key information to help you decide whether to participate. Detailed information follows this brief summary. Ask the research team questions. Taking part in this study is completely voluntary.

#### WHAT IS THE STUDY ABOUT AND HOW LONG WILL IT LAST?

The purpose of this research is to understand the experiences and health outcomes of veterans who get legal services in different settings. This research project is a clinical trial. Half of the participants will be assigned to get their legal help from the Connecticut Veterans Legal Center (CVLC), and half will get it from state groups in the community. CVLC is a legal center based at VA Connecticut. Whether you are assigned to CVLC or legal help in the community will be determined by chance (like a coin flip), with a 50% chance of getting each type of legal help. Your participation in this research will last about 12 months.

If you decide to participate, you will complete four interviews with a research assistant. During the first interview, you will be asked questions about your background, physical and mental health, substance use, housing, income, and legal problems you may be experiencing. Follow-up interviews will be scheduled about 3 months, 6 months, and 12 months after the first interview and will include similar questions.

Information about your health, diagnoses, and use of VA services will be provided to us by the VA Connecticut Healthcare System (VACHS). If you receive legal services from the Connecticut Veterans Legal Center (CVLC), information about the legal services you received will be provided to us for research purposes.

You may be asked to complete two additional interviews with a research staff member 3 months and 6 months after your first interview. The purpose of these interviews is to learn more about your experience getting legal services and how your legal situation is impacting your life. These discussions will be audio-recorded.

We will ask you for the name and contact information of three people who will be able to help us get in touch with you for study assessments in case we cannot reach you at the number you provide. You should inform these people that you are in a research study and that someone from our team may call them in case you cannot be reached. We will not share any information with these contact people except that you are participating in a research study.

#### WHAT ARE KEY REASONS YOU MIGHT CHOOSE TO VOLUNTEER FOR THIS STUDY?

### RESEARCH CONSENT FORM

# **VA Connecticut Healthcare System**

| Subject Name: | Date: |
|---|---|
| Title of Study: Medical-legal partnerships to prevent evictions and homelessn | ess among veterans |
| Principal Investigator: Marc Rosen, M.D. | Version Date: v.04/05/2023 |

You will not be directly helped by taking part in this study. However, your participation may lead to knowledge that will help others. Results of this project may help us understand how providing legal services to veterans can impact their health and their lives.

Participation in any part of the project will not delay or modify any services you are eligible to receive from the CVLC or the VA Healthcare System. Regardless of study participation, you are allowed to request CVLC services at any time. No extra services will be provided because you are participating in this project. It is unlikely, but if there is a waitlist for CVLC services, you may get CVLC services sooner if you are assigned to the CVLC group.

# WHAT ARE KEY REASONS YOU MIGHT CHOOSE NOT TO VOLUNTEER FOR THIS STUDY?

Answering survey questions takes time you may not want to spend (although you will be paid for the time you spend completing the surveys). There is a risk that answering questions about your legal problems, mental health, substance use, or life may be upsetting. There is also a very small risk that the information you provide could be revealed to someone outside of this research project. However, steps will be taken to keep your information from being revealed outside this project.

## DO YOU HAVE TO TAKE PART IN THE STUDY?

If you decide to take part in the study, it should be because you really want to volunteer. You will not lose any services, benefits, or rights you would normally have if you choose not to volunteer.

#### **RESEARCH DETAILS**

# WHAT IS THE PURPOSE OF THIS STUDY?

By conducting this research study, we hope to learn about how legal services offered in different settings impact health outcomes and veterans' housing situations. We also hope to better understand how legal providers can best help veterans.

## HOW LONG WILL YOU BE IN THE STUDY?

This research study is expected to take about four years. Your individual participation in the project will last 12 months.

### RESEARCH CONSENT FORM

# **VA Connecticut Healthcare System**

| Subject Name: | Date: |
|---|---|
| Title of Study: Medical-legal partnerships to prevent evictions and homelessness among veterans | |
| Principal Investigator: Marc Rosen, M.D. | Version Date: v.04/05/2023 |

#### WHAT WILL HAPPEN IF YOU TAKE PART IN THE STUDY?

If you choose to participate in this study, this is what will happen. First, you will be interviewed by a research assistant. During this interview, you will be asked questions about your background, physical and mental health, substance use, housing, income, and legal problems you may be experiencing. We will also ask you to provide the name and contact information of three people who can help us get in touch with you for follow-up interviews in case we cannot reach you. This first interview will take about one hour to complete. After that interview, you will be assigned by chance (like a flip of a coin) to receive your legal services from CVLC or from pro-bono legal providers in the community.

If you are assigned to get services from CVLC, your CVLC legal providers will communicate with your VA Connecticut healthcare providers and share relevant health and legal information with each other.

If you are assigned to the group that gets legal services in the community, you will be given the phone number and/or website of the agency in the community that helps people being evicted with their legal problems.

After your first interview, you will have three more interviews with the research assistant scheduled 3 months, 6 months, and 12 months after the first interview. Questions for each of these follow-up interviews will be similar to those you completed in the first interview. Each follow-up interview will take about 45 minutes to complete.

Approximately 30 participants will be asked to complete two additional interviews with the study team. If you are part of this group, you will be interviewed 3 months and 6 months after your first interview. Unlike your first interview, this interview will be recorded, and you will be asked about your experiences with legal providers, and how your legal situation is impacting your life. These discussions will take about 30 minutes to complete.

#### WHAT IS EXPECTED OF YOU IF YOU TAKE PART IN THIS STUDY?

If you decide to participate in this research study, please:

- Keep your study appointments. If you miss an appointment, please contact the research staff to reschedule as soon as you know you will miss the appointment.
- Answer questions as instructed and ask questions as you think of them so that you can
  give your best answer. You can refuse to answer any questions that you don't want to
  answer. It is better to refuse than to answer is a way that is not accurate.

# WHAT POSSIBLE RISKS OR DISCOMFORTS MIGHT YOU HAVE IF YOU TAKE PART IN THIS STUDY?

Any procedure has possible risks and discomforts. The procedures in this study involve answering questions about yourself in an interview. Some people become uncomfortable or

### RESEARCH CONSENT FORM

# **VA Connecticut Healthcare System**

| Subject Name: | Date: |
|---|---|
| Title of Study: Medical-legal partnerships to prevent evictions and homelessness among veterans | |
| Principal Investigator: Marc Rosen, M.D. | Version Date: v.04/05/2023 |

upset at being asked questions about their legal problems, housing situation, health, or substance use. You can skip any questions that you do not want to answer for any reason, and you can stop the interview if you want to. Another risk of participating in this project is that information you share might become known to other people outside of the research team. To minimize this risk, we will take steps to keep your information safe.

Risks of the usual care you receive at VA Connecticut, CVLC, or from other legal providers in the community are not risks of this study. Those risks are not included in this consent form. You should talk with your healthcare and legal providers if you have any questions about the risks of these services.

#### WHAT ARE THE POSSIBLE BENEFITS OF THIS STUDY?

If you are assigned to get legal services at CVLC and there is a waiting list for getting services, participation in this study will get you those services faster. That is unusual – usually there is no waiting list for CVLC services. If there is no waitlist for getting services from CVLC or you are assigned to receive legal services in the community, you will not be directly helped by taking part in this study but your participation may lead to knowledge that may help others like you who are facing similar legal problems.

# WHAT OTHER CHOICES DO YOU HAVE IF YOU DO NOT WANT TO JOIN THIS STUDY?

You may choose not to participate in this study. If this is your decision, you can still get legal services from CVLC or ask CVLC for a referral to legal services in the community. Participation in this study is completely voluntary and if you withdraw from the research project, your withdrawal will not affect your ability to get services you are eligible for from CVLC, community legal services, or the VA Connecticut Healthcare System.

# **HOW WILL YOUR PRIVATE INFORMATION BE PROTECTED?**

Taking part in this study will involve collecting private information about you. This information will be protected in the following ways:

- All paper records will be stored in a locked filing cabinet in a locked research office.
- All electronic records will be stored on a password-protected computer that is behind the VA firewall.
- Only authorized research staff will have access to paper and electronic research records.
- The information collected from this study will be kept separate from your name and contact information. The data will be coded with a random code number that cannot be used to identify you. The master file linking your name to the code number will be kept separate and will only be accessible by the research staff.
- Your name or identifying information will not be revealed in any reports or publications resulting from this study.

### RESEARCH CONSENT FORM

# **VA Connecticut Healthcare System**

| Subject Name: | Date: |
|---|---|
| Title of Study: Medical-legal partnerships to prevent evictions and homelessness among veterans | |
| Principal Investigator: Marc Rosen, M.D. | Version Date: v.04/05/2023 |

There are times when we might have to show your records to other people. For example, our local Research and Development Committee, VA officials, or other study monitors may look at or copy portions of records that identify you.

Identifiers might be removed from your private information that is collected. After that removal, the information could be used for future research studies or distributed to another investigator for future research studies without additional informed consent from you or your legally authorized representative.

We will include information about your study participation in your VA medical record if you have one. A note will be added stating that you are participating in this study. Information collected from study interviews will not be included in that note. Federal laws and regulation that protect privacy of medical records will apply to your VA record.

A description of this clinical trial will be available on a website called ClinicalTrials.gov as required by U.S. Law. This website will not include information that can identify you. At most, the website will include a summary of the results of this study. You can search this website at any time.

# WHAT ARE THE COSTS TO YOU IF YOU TAKE PART IN THIS STUDY?

You will not be charged for any treatments or procedures that are part of this study. If you usually pay co-payments for VA care and medications, you will still pay these co-payments for VA care and medications that are not part of this study.

## IS THERE PAYMENT TO YOU IF YOU TAKE PART IN THIS STUDY?

You will be paid for participating in this study as follows, for a total of up to \$180:

- First interview (Baseline) with research assistant: \$40
- Second interview (3-month follow-up) with research assistant: \$40
- Third interview (6-month follow-up) with research assistant: \$50
- Fourth interview (12-month follow-up) with research assistant: \$50

If you are selected to be in the small group that completes additional, recorded interviews asking about experiences of legal services, you will be paid as follows, for up to an additional \$60:

3-month interview: \$30 6-month interview: \$30

Payment will be issued after each assessment is completed by secure electronic transfer from the VA to your bank account or by a check mailed to your home address.

#### WHAT WILL HAPPEN IF YOU ARE INJURED BECAUSE OF YOUR BEING IN THE STUDY?

#### RESEARCH CONSENT FORM

# **VA Connecticut Healthcare System**

| Subject Name: | Date: |
|---|---|
| Title of Study: Medical-legal partnerships to prevent evictions and homelessness among veterans | |
| Principal Investigator: Marc Rosen, M.D. | Version Date: v.04/05/2023 |

If you are injured as a direct result of your participation in this research study, VA will provide necessary medical treatment at no cost to you. Emergency and ongoing medical treatment will be provided as needed. Except in very limited circumstances, this medical treatment will be provided in a VA Medical facility. There are no plans to provide compensation for disability or other losses occurring over the long term or if an injury becomes apparent after your participation in the study has ended. However, by agreeing to participate in this research study, you are not waiving or giving up any legal rights to seek compensation.

If you should have a medical concern or get hurt or sick as a result of taking part in this study, call:

 The VA Connecticut Human Studies Research Coordinator at 1-203-937-3830

OR

• The study Principal Investigator, Dr. Marc Rosen at 1-203-932-5711 x1-2112

#### WHO ELSE MAY YOU CONTACT IF YOU HAVE QUESTIONS?

If you have questions about your rights as a study subject, or you want to make sure this is a valid VA study, you may contact the Chairman of the Human Studies Subcommittee at 1-203-932-5711 x1-3350.

If you have questions, complaints or concerns about the study or if you would like to obtain information or offer input you may call the study Principal Investigator, Dr. Marc Rosen at 1-203-932-5711 x1-2112.

#### DO YOU HAVE TO TAKE PART IN THE STUDY?

Participation in this study is completely voluntary and your decision to participate or withdraw from the research project will involve no penalty or loss of benefits to which you are otherwise entitled and will not affect services you receive from CVLC or the VA Connecticut Healthcare System.

## RIGHT OF INVESTIGATOR TO TERMINATE YOUR PARTICIPATION

The research staff might end your participation in this study if you are rude or threatening to staff, or in some other way are judged unable to safely complete study participation.

# RESEARCH CONSENT FORM

# **VA Connecticut Healthcare System**

| Subject Name: | | Date: |
|---|---|---|
| Title of Study: Medical-legal partn | erships to prevent evictions and homele | ssness among veterans |
| Principal Investigator: Marc Rose | en, M.D. | Version Date: v.04/05/2023 |
| AGREEMENT TO PARTICIPATE IN THE RESEARCH STUDY | | |
| You have been told of the risl been told of other choices of ask questions and obtain ans By signing this document beloconfirm that you have read the a copy of this consent document | ow, you voluntarily consent to participate | of the study. You have sen given the chance to sen this study You also d to you. You will receive |
| Subject's Name | Subject's Signature | Date |
| Person Obtaining Consent | Person Obtaining: Signature | <br>Date |